CLINICAL TRIAL: NCT05182255
Title: Post Market Clinical Study - Evolution® Esophageal Stent Systems, Europe: Fully and Partially Covered
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: MDR-2054
Record Dates: First submitted 2021-12-16; First posted 2022-01-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Diseases
Keywords: Unresectable esophageal malignancies; Benign strictures; Tracheoesophageal fistulas; Esophageal stents
MeSH Terms: conditions — Esophageal Diseases; Tracheoesophageal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Esophageal Stent Systems: Freedom from endoscopic re-intervention due to recurrence of dysphagia
  Interventions: Device: Evolution® Esophageal Stent Systems, Europe: Fully and Partially Covered

INTERVENTIONS:
Device: Evolution® Esophageal Stent Systems, Europe: Fully and Partially Covered — To aid in maintaining patency of the esophagus in cases of obstruction of the esophagus caused by an esophageal disease and to seal tracheoesophageal fistula.

SUMMARY:
The aim of this post-market clinical follow-up study is to evaluate the continued safety and performance of the marketed Evolution® Esophageal Stent System (Partially- and Fully Covered).

DETAILED DESCRIPTION:
Cook Evolution® Esophageal Stent Post-Market Data Collection Study

A retrospective observational, multi-center, chart review study will be performed. Data specific to Cook Evolution® Esophageal Stent placement procedures from all consecutive patients who underwent stent placement with any of the stents at the participating sites between 1st January 2015 and 31st December 2020 (index period) will be collected. Research on the commercially available Cook Evolution® Esophageal Stents is being conducted to comply with the new medical device regulation, EU 2017/745, to assess the device for its continued safety and performance. To do this, Cook Research Incorporated is working with participating hospitals to collect pseudonymized (coded) personal health data. This study is in the interest of public health; to learn more about the necessary data processing, please visit the webpage below.

https://www.cookresearchinc.com/extranet/pdf/2054-55_Data_Protection_Notice.pdf

Spanish: https://www.cookresearchinc.com/extranet/pdf/2054-55_Data_Protection_Notice_ESP.pdf

ELIGIBILITY:
Inclusion Criteria:

1: Patient has had at least one of the following stents implanted between 1st January 2018 and 31st December 2020*:

* Evolution® Esophageal Stent System-Partially Covered
* Evolution® Esophageal Stent System-Fully Covered
* Evolution® Esophageal Stent System-Fully Covered

Exclusion Criteria:

1: Deceased retrospective patient who has set post-mortem instruction against processing of his/her health data

2. Patient or his/her legally authorized representative objects to collection and processing of his/her data, or not willing to sign not willing to sign an Informed consent, if it is required by the local EC committee. There may be local exemptions where consent is not a requirement or non-objection letters may replace informed consent processes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who underwent stent placement with a study device between Jan 1,2018 thru Dec 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically relevant device migration | 6 months
  Clinically relevant device migration is defined as stent migration requiring replacement of the stent due to degree of migration as well as clinical symptoms (i.e. an inability of the stent to perform its intended function).

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (3):
  - Klinikum Altenburg, Altenburg
  - Universitatsklinikum Augsburg, Augsburg
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
- Hospital Universitario de Salamanca, Salamanca, ESP, Spain
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after final report has been distributed and ending 5 years after final report has been distributed. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.